CLINICAL TRIAL: NCT07362368
Title: Validity and Reliability of the Immersive Virtual Reality Adaptation of the Five-Repetition Sit-to- Stand Test in Asymptomatic Young Adults
Brief Title: Virtual Reality-Based Five-Repetition Sit-to-Stand Test in Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_VR5STS_ADAPTATION_1
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Functional Mobility; Virtual Reality-Based Functional Assessment
Keywords: Functional Mobility; Five-Repetition Sit-to-Stand Test; Virtual Reality; Immersive Virtual Reality; Validity; Reliability; Young Adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic Young Adults: Asymptomatic young adults aged 18-30 years undergoing conventional and immersive virtual reality-based Five-Repetition Sit-to-Stand assessments to evaluate feasibility, validity, and reliability.
  Interventions: Other: Clinical Assessments

INTERVENTIONS:
Other: Clinical Assessments — Participants will perform the Five-Repetition Sit-to-Stand test using an immersive virtual reality application developed for the Meta Quest 3 platform. The virtual environment digitally replicates the conventional test setup, including chair height, starting position, movement sequence, and completion criteria. Test duration will be automatically recorded by the system. The virtual reality-based assessment is designed to provide a standardized, objective, and reproducible evaluation of lower extremity functional performance and will be repeated to assess test-retest reliability.

SUMMARY:
Lower extremity muscle strength is a fundamental determinant of an individual's ability to maintain functional mobility, preserve balance, and perform activities of daily living independently. One of the methods used for the comprehensive evaluation of these functions is the Five-Repetition Sit-to-Stand (5STS) test, which is considered an effective tool for assessing lower extremity strength, balance, and functional mobility in both healthy individuals and various clinical populations. In this test, participants are required to consecutively stand up from and sit down on a chair five times without using their arms, and the completion time is recorded in seconds to objectively evaluate functional capacity. Due to its simplicity, low cost, and high reliability, the 5STS test is widely used in clinical and research settings.

However, functional tests administered in conventional clinical environments may be insufficiently standardized due to factors such as examiner-related variability, measurement errors, and environmental influences. This limitation makes it difficult to detect small performance differences and restricts test repeatability. In recent years, rapidly advancing virtual reality (VR) technology has contributed to overcoming these limitations by offering the potential to digitally standardize measurement processes. VR systems, which recreate real-life scenarios in a three-dimensional and interactive manner, allow for a more comprehensive and objective assessment of motor performance. In addition, by increasing user interaction and reducing observer-related errors, VR enhances clinical validity. One study has reported that the most important advantage of VR in clinical balance assessments is its ability to provide a fully controllable, repeatable, and standardized environment. Similarly, a systematic review found that VR-based exercises resulted in significant improvements in motor skills, balance, and cognitive function, while increasing user engagement and motivation and thereby contributing to more effective rehabilitation outcomes.

Current literature indicates that VR technology is increasingly being utilized in physiotherapy and exercise sciences. In one study, the validity and feasibility of a VR adaptation of the Wingate Anaerobic Test were investigated, and it was reported that the VR version produced performance outcomes comparable to the conventional test, while participant satisfaction was significantly higher with the VR-based method. Likewise, another study demonstrated that the VR adaptation of the Six-Minute Pegboard and Ring Test exhibited high levels of validity and reliability. Together, these studies indicate that VR-based functional tests are both feasible and clinically consistent.

Despite this, no studies to date have examined the validity and reliability of the Five-Repetition Sit-to-Stand test in an immersive VR environment for assessing lower extremity function. Therefore, the present study aims to determine the validity, reliability, and feasibility of a virtual reality-based Five-Repetition Sit-to-Stand test (5STS-VR) developed on the Meta Quest 3 platform in asymptomatic young adults. Additionally, convergent validity will be evaluated by analyzing the relationships between performance data obtained from the virtual environment and outcomes of the Y-Balance Test and lower extremity muscle strength measurements.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years,
* Asymptomatic, with no neurological, cardiovascular, or musculoskeletal symptoms,
* Ability to perform activities of daily living independently,
* Visual, auditory, and vestibular functions adequate for virtual reality applications,
* Ability to understand and follow instructions in Turkish,
* Willingness to participate voluntarily in the study.

Exclusion Criteria:

* History of lower extremity injury, surgical procedure, or serious musculoskeletal condition within the past six months,
* Presence of vestibular disorders, balance impairment, or visual or hearing impairments,
* Experiencing symptoms of VR sickness, such as dizziness, nausea, or spatial disorientation during virtual reality applications,
* Diagnosis of neurological, cardiovascular, or metabolic disease,
* Engaging in intensive exercise or being a professional athlete,
* Insufficient cognitive ability to understand test instructions,
* Voluntary withdrawal from the study during the research process.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic young adults aged 18-30 years who are able to perform activities of daily living independently and have no neurological, cardiovascular, or musculoskeletal conditions affecting functional performance.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Five-Repetition Sit-to-Stand Test - Virtual Reality (5STS-VR) | Baseline and 1-week follow-up
  This outcome measure will be used to assess lower extremity functional performance using an immersive virtual reality-based adaptation of the Five-Repetition Sit-to-Stand test. Test completion time will be automatically recorded by the system. Validity will be evaluated by comparison with the conventional Five-Repetition Sit-to-Stand test, and reliability will be assessed using repeated measurements performed one week apart.

SECONDARY OUTCOMES:
Five-Repetition Sit-to-Stand Test - Conventional | Baseline
  The conventional Five-Repetition Sit-to-Stand test will be administered to assess lower extremity strength and functional mobility and will be used as a reference measure for concurrent validity analysis.
Y-Balance Test | Baseline
  The Y-Balance Test will be used to assess dynamic balance and postural control. Results will be used to examine convergent validity of the virtual reality-based Five-Repetition Sit-to-Stand test.
Lower Extremity Muscle Strength | Baseline
  Lower extremity muscle strength will be measured using a handheld digital dynamometer to evaluate its relationship with functional performance and virtual reality-based Five-Repetition Sit-to-Stand outcomes.
Participant Satisfaction | Baseline
  Participant satisfaction with conventional and virtual reality-based assessments will be evaluated using a 10-point visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Yusuf ÖZBAĞ, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maden C, Gozacan Karabulut D, Bagci B. Validity and reliability of an immersive virtual reality adaptation of the 6-minute pegboard and ring test. Hand Surg Rehabil. 2025 Feb;44(1):101981. doi: 10.1016/j.hansur.2024.101981. Epub 2024 Oct 30. PMID 39486588
- [Background] Bayram GA, Sahin GE, Yilmaz G, Tayboga UI, Celik AG, Yildirim Y, Saribas PK, Tarakci D. Integration of the wingate anaerobic test into a virtual reality- based evaluation system. BMC Sports Sci Med Rehabil. 2025 Jul 2;17(1):163. doi: 10.1186/s13102-025-01220-4. PMID 40605090
- [Background] Ali SG, Wang X, Li P, Jung Y, Bi L, Kim J, Chen Y, Feng DD, Magnenat Thalmann N, Wang J, Sheng B. A systematic review: Virtual-reality-based techniques for human exercises and health improvement. Front Public Health. 2023 Mar 23;11:1143947. doi: 10.3389/fpubh.2023.1143947. eCollection 2023. PMID 37033028
- [Background] Morel M, Bideau B, Lardy J, Kulpa R. Advantages and limitations of virtual reality for balance assessment and rehabilitation. Neurophysiol Clin. 2015 Nov;45(4-5):315-26. doi: 10.1016/j.neucli.2015.09.007. Epub 2015 Oct 31. PMID 26527045
- [Background] Scott H, Griffin C, Coggins W, Elberson B, Abdeldayem M, Virmani T, Larson-Prior LJ, Petersen E. Virtual Reality in the Neurosciences: Current Practice and Future Directions. Front Surg. 2022 Feb 18;8:807195. doi: 10.3389/fsurg.2021.807195. eCollection 2021. PMID 35252318
- [Background] Rizzo AS, Koenig ST. Is clinical virtual reality ready for primetime? Neuropsychology. 2017 Nov;31(8):877-899. doi: 10.1037/neu0000405. PMID 29376669
- [Background] Munoz-Bermejo L, Adsuar JC, Mendoza-Munoz M, Barrios-Fernandez S, Garcia-Gordillo MA, Perez-Gomez J, Carlos-Vivas J. Test-Retest Reliability of Five Times Sit to Stand Test (FTSST) in Adults: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Jun 9;10(6):510. doi: 10.3390/biology10060510. PMID 34207604